CLINICAL TRIAL: NCT06911060
Title: The Effect of Flaxseed Consumption on Biochemical Parameters and Quality of Life in Patients With Type 2 Diabetes
Brief Title: Flaxseed Consumption on Biochemical and Quality of Life in Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, YASEMİN ERTAŞ ÖZTÜRK, Assist. Prof., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BAP08-2025-5797; BAP08-2025-5797 (Other Grant/Funding Number: Ondokuz Mayıs University Scientific Research Project)
Record Dates: First submitted 2025-03-12; First posted 2025-04-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 diabetes mellitus; flaxseed; quality of life; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linseed Oil; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet+Flaxseed (Experimental): Diet will be planned to patients with T2DM as a part of their medical nutritional therapy. This group will take 30 g/d ground flaxseed within their diet.
  Interventions: Dietary Supplement: Flaxseed; Behavioral: Diet
- Diet (Experimental): Diet will be planned to patients with T2DM as a part of their medical nutritional therapy.
  Interventions: Behavioral: Diet

INTERVENTIONS:
Dietary Supplement: Flaxseed — 30 g/day for 12 weeks
  Arms: Diet+Flaxseed
Behavioral: Diet — Diet will be planned to patients with T2DM as a part of their medical nutrition therapy.

SUMMARY:
The main goal of this clinical trial is to determine the effect of flaxseed added to the diet on biochemical parameters and quality of life in patients with Type 2 diabetes mellitus (T2DM). The main questions it aims to answer are:

* Does flaxseed supplementation given to T2DM patients for 12 weeks have an effect on biochemical parameters?
* Does flaxseed supplementation given to T2DM patients for 12 weeks have an effect on quality of life?

Researchers will compare patients with T2DM consume diet added flaxseed to a control group to see if flaxseed effect on biochemical parameters and quality of life.

Participants will:

* Complete the questionnaire, record the 3-day food consumption and be taken the anthropometric measurements at the beginning and end of the study.
* Take diet added 30 g ground flaxseed (intervention group) or only diet (control group) every day for 12 weeks.
* Visit the clinic once every 4 weeks for follow-up.
* Report the dietary adherence and gastrointestinal symptoms on a phone call once every week.

DETAILED DESCRIPTION:
Adult individuals between the ages of 19-65, with a body mass index (BMI) between 20-35 kg/m2, using oral anti-diabetics and not using insulin will be included in the study. Patients with T2DM who agree to participate in the study will be randomly assigned to the intervention or control group using the simple randomization method. Participants will be followed for 12 weeks. Both groups will receive diet as part of T2DM treatment. Subjects in the intervention group will consume 30 g of ground flaxseed per day in addition to their diet. The participants were asked by the researchers through a face-to-face interview technique to determine their demographic characteristics (age, marital status, education level, employment status, income level, etc.), quality of life short form (SF-36) scale, international physical activity questionnaire (IPAQ) and 3-day food consumption record. A survey form questioning consumption records will be applied at the baseline and end of the study. In addition, routinely monitored biochemical parameters of the patients will be recorded from the hospital system at the baseline and end of the study. Anthometric measurements will be taken and recorded by the researcher in accordance with the method. The data obtained will be evaluated in the SPSS package program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2DM by a physician
* Being between the ages of 19-65
* Having a body mass index (BMI) between 20-35 kg/m2
* Using oral anti-diabetics and not using insulin

Exclusion Criteria:

* History of gastrointestinal diseases
* High consumption of nuts, flaxseeds or sesame seeds (more than one serving per day)
* Food allergies or intolerances
* Malignancies
* Renal failure, liver, other endocrine or inflammatory disorders
* Use of lipid-lowering drugs
* Smoking and alcohol use
* Being pregnant or lactating

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of flaxseed on fasting blood glucose (mg/dL) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on HbA1c (%) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on total triglyceride (mg/dL) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on total cholesterol (mg/dL) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on HDL-cholesterol (mg/dL) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on LDL-cholesterol (mg/dL) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on quality of life | From enrollment to the end of intervention at 12 weeks
  Quality of life will be assessed with SF-36. The total score is evaluated separately into two summary scores: the physical component summary (PCS12) and the mental component summary (MCS12). The score of the answers related to the PCS12 is obtained from the factors of general health, role-physical, physical functioning, and bodily pain, and the score of the answers related to the MCS12 is obtained from the factors of social functioning, role-emotional, mental health, and energy/fatigue. Both scores range from 0 to 100, with a higher score representing better health.

SECONDARY OUTCOMES:
Evaluation of the effect of flaxseed on BMI (kg/m2) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on waist circumference (cm) | From enrollment to the end of intervention at 12 weeks
Evaluation of the effect of flaxseed on waist/hip ratio | From enrollment to the end of intervention at 12 weeks